CLINICAL TRIAL: NCT00348153
Title: Randomized Controlled Study to Evaluate the Efficacy of Adalimumab in Patients With Different Forms of Refractory Uveitis Acronym: Adalimumab in Uveitis Refractory to Conventional Therapy (ADUR Trial)
Brief Title: Adalimumab in Uveitis Refractory to Conventional Therapy (ADUR Trial)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heidelberg University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Friederike Mackensen, PD Dr. med., Heidelberg University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT: 2006-001732-53
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Uveitis
Keywords: Uveitis; Adalimumab; TNF alpha
MeSH Terms: conditions — Uveitis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Adalimumab + corticosteroids + immunosuppressive treatments (Experimental): Adalimumab 40 mg eow, stable immunosuppression, corticosteroids in 1 mg/kg/Bodyweight (max. 80 mg) and taper
  Interventions: Drug: Adalimumab
- immunosuppressive treatment + corticosteroids (Active Comparator): corticosteroids upped to 1mg/kg/Bodyweight and taper, stable immunosuppressive treatment
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab

SUMMARY:
TNF alpha Inhibitors have been very effective in treating rheumatologic diseases as well as uveitis. Adalimumab is the first member of a new class of TNF antibody compounds developed to contain exclusively human sequences. We want to test the efficacy and safety of the TNF alpha Inhibitor Adalimumab in patients with active uveitis despite standard immunosuppressive therapy.

DETAILED DESCRIPTION:
TNF alpha Inhibitors like Infliximab and Etanercept have been very effective in treating rheumatologic diseases. They have been used to treat severe uveitis by several groups, Suhler and coworkers have published the largest series in 2005. Adalimumab, a recombinant, full-length immunoglobulin, is the first member of a new class of TNF antibody compounds developed to contain exclusively human sequences. The duration of therapeutic efficacy of other TNF antibodies, which contain non-human sequences, may be limited to a greater extent by antibody responses raised in subjects over time. We want to test the efficacy and safety of the TNF alpha Inhibitor Adalimumab in patients with active uveitis despite standard immunosuppressive therapy requiring systemic corticosteroids > 7,5mg prednisolone.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 18 and older
* Subjects must meet the criteria for non-infectious uveitis according to the definition of the SUN working group
* Uveitis must have first been diagnosed at least 6 months ago
* Persistence of active disease ( > 2 flares within 6 months) or progressive deterioration of vision (< 0,6) within the last 3 months despite immunosuppressive therapy requiring corticosteroids ≥ 7,5 mg prednisone
* Women of childbearing potential have to practice a reliable birth control method throughout the study and until five months after the last administration of Adalimumab
* Ability to comprehend and willing to give informed consent for participation in the study
* Able and willing to self-administer sc injections or assistance of a suitable person to administer sc injections
* Negative PPD skin test or serological testing according to official German recommendations for tuberculosis testing AND chest X-ray within the last three month. Treatment of latent TB with INH must be started 4 weeks prior to administration of first dose of study drug.

Exclusion Criteria:

* Participation in another clinical trial and/or observation period of competing trials
* Treatment with infliximab within the last 2 months or with etanercept within the last 3 weeks
* Patients with only intermediary uveitis or optic neuritis multiple sclerosis
* Patients with uveitis caused by infection
* Patients with optic atrophy, macular scar, cataract, amblyopia or corneal scars
* Patients with recurrent episodes of uveitis, but long intermittent phases of complete remissions without therapy
* Patients possibly demanding vitrectomy or cataract surgery within the time of clinical trial
* Pregnant and nursing women or women planning a pregnancy within 5 months
* Persistent or recurrent infections or severe infections requiring hospitalization with iv antibiotics within 30 days, or oral antibiotics within 14 days prior to enrollment
* Known opportunistic infection (such as herpes zoster) during the last 2 months
* Live vaccination during the last 30 days
* History of tuberculosis; histoplasmosis or listeriosis
* Known HIV infection, active hepatitis B or C
* Comorbidities: uncontrolled diabetes, unstable ischemic heart disease, congestive heart failure (NYHA III, IV), active inflammatory bowl disease, recent stroke (within three months), chronic leg ulcer and similar conditions which would put the subject at risk by participation in the trial
* Previous diagnosis of signs of central nervous system demyelinating diseases
* History of cancer or lymphoproliferative disease other than a successfully and completely treated squamous cell or basal cell carcinoma of the skin or cervical dysplasia, with no recurrence within the last two years
* Hemoglobin < 10 g/dl, white blood cell count < 3.0x109/l, platelet count < 100x109/l, creatinine level >1.5 mg/dl, liver enzymes > 1.5 times above normal or alkaline phosphatase >3 times above normal
* Clinical examination showing significant abnormalities of clinical relevance
* Current evidence of significant abuse of drugs
* Psychiatric disease/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-08; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Improvement of visual acuity (3 lines EDTRS) | at week 0, 2, 6, 12 and 24

SECONDARY OUTCOMES:
Improvement of intraocular inflammatory activity | at week 0, 2, 6, 12 and 24
Evolution of cystoid macula edema(FLA, OCT) | at week 0, 6, 12 and 24
Number of switchers from Arm A to Arm B | after six months
Cumulative steroid dosage | after six months
Frequency of adverse events | whole study period

CONTACTS AND LOCATIONS:
Overall Officials: Hannes M Lorenz, MD, Principal Investigator — Department of Rheumatology, University of Heidelberg; Matthias D Becker, MD, Principal Investigator — Interdisziplinary Uveitis Center, University of Heidelberg; Regina Max, MD, Study Director — Interdisziplinary Uveitis Center, University of Heidelberg
Locations (1):
- Interdisciplinary Uveitis Center, University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Becker MD, Smith JR, Max R, Fiehn C. Management of sight-threatening uveitis: new therapeutic options. Drugs. 2005;65(4):497-519. doi: 10.2165/00003495-200565040-00005. PMID 15733012
- [Background] Lim L, Suhler EB, Smith JR. Biologic therapies for inflammatory eye disease. Clin Exp Ophthalmol. 2006 May-Jun;34(4):365-74. doi: 10.1111/j.1442-9071.2006.01225.x. PMID 16764659
- [Background] Suhler EB, Smith JR, Wertheim MS, Lauer AK, Kurz DE, Pickard TD, Rosenbaum JT. A prospective trial of infliximab therapy for refractory uveitis: preliminary safety and efficacy outcomes. Arch Ophthalmol. 2005 Jul;123(7):903-12. doi: 10.1001/archopht.123.7.903. PMID 16009830
- [Background] Smith JR, Levinson RD, Holland GN, Jabs DA, Robinson MR, Whitcup SM, Rosenbaum JT. Differential efficacy of tumor necrosis factor inhibition in the management of inflammatory eye disease and associated rheumatic disease. Arthritis Rheum. 2001 Jun;45(3):252-7. doi: 10.1002/1529-0131(200106)45:33.0.CO;2-5. PMID 11409666